CLINICAL TRIAL: NCT02220881
Title: Effectiveness of Mold Making Silicone Toe Separator on Hallux Valgus: A Prospective, Randomized Single-Blinded Controlled Trial
Brief Title: Mold Making Silicone Toe Separator on Hallux Valgus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Navaporn Chadchavalpanichaya, Assistance Professor, Mahidol University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: silicone HV
Record Dates: First submitted 2014-01-08; First posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Hallux Valgus
Keywords: Hallux valgus, Mold making silicone toe separator, Toe separator
MeSH Terms: conditions — Hallux Valgus | interventions — Observation; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mold making silicone toe separator (Experimental): The subject in experimental group will use mold making silicone toe separator everyday
  Interventions: Device: Mold making silicone toe separator
- Observation (Other): This group will follow the physician instruction of care for the hallux valgus
  Interventions: Other: Observation

INTERVENTIONS:
Device: Mold making silicone toe separator — Each subject in the controlled receives the custom-made mold making silicone toe separator made by certified orthotist and the recommendation of use the proper shoes without determination of current drug use
  Other Names: Toe separator
  Arms: Mold making silicone toe separator
Other: Observation — The participants in this groups will be educated on how to care the hallux valgus without any intervention. The follow up will be on the 3rd, 6th, 9th and 12th month.
  Other Names: Control group
  Arms: Observation

SUMMARY:
The primary objective of this study is to investigate the effectiveness of mold making silicone toe separator on reducing the hallux valgus angle. In addition, this study aims to determine the compliance of mold making silicone toe separator, the change in pain level and, including, the satisfaction of the participants after using mold making silicone toe separator.

DETAILED DESCRIPTION:
Study Protocol, Data collection

Ninety recruited sample is the patient come to the foot clinic, Siriraj Hospital with the age over eighteen years old, presence of hallux valgus deformity in moderate level (without the condition of hallux rigidus), and never use hallux valgus strap or toes separator before.

The sample is given a physical assessment by physician and is asked to fill in a self-administered questionnaire which composes of general information, the foot problem information and the impact of deformity to patients function information. General information section requires the detail regarding age, genders, and the average walking hours. Foot problem information section composes of side, duration of hallux valgus and family history. Impacts of the hallux valgus deformity section includes walking problem, shoes-fitting problem, working problem, and daily activities problem, were recorded by using a numeric rating scale from 0 to 10; 0 refers as no problem and 10 refers as the worst problem. The sample then will be taken the radiograph of the feet in order to evaluate the degree of hallux valgus angle and intermetatarsal angle.

After the completion of assessment, the sample is randomly divided into 2 groups; control and experimental group by using computer program.

* Control group receives the recommendation of use the proper shoes without determination of current drug use
* Experimental group receives the custom-made mold making silicone toe separator made by certified orthotist and the recommendation of use the proper shoes without determination of current drug use

The follow up activity is on every 3rd, 6th, 9th and 12th of the study period in both groups by using questionnaire; pain score (NRS), satisfaction of using the custom-made mold making silicone toe separator (NRS) and report of complication. In the 6th and 12th month, the progress evaluation on hallux valgus and intermetatarsal angle is done by radiograph. The angle then is recorded by mean of the three values.

Descriptive statistics; mean, standard deviation or interquartile range, will be used to identify the demographic data of the participant and compliance of device usage. Analytical statistics; Unpaired t-test or Mann Whitney U test will be used for determining the average device usage time, pain score, and satisfaction of the participants after using mold making silicone toe separator.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years of age
* Presence of hallux valgus deformity in moderate level, if the condition presents in both side, the one with greater angle will be selected
* Never use hallux valgus strap or toes separator before

Exclusion Criteria:

* Presence of hallux rigidus and hallux limitus
* Presence of acute hallux inflammation
* Experience the use hallux valgus strap or toes separator in a past year
* Experience the allergy to silicone

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-06 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of degree of Hallux valgus angle at month 6 ans month 12 | Baseline, month 6, month 12
  Hallux valgus angle will be measured from the x-ray film taken in standing position with full weight bearing
Change from baseline of degree of intermetatarsal angle at month 6 ans month 12 | Baseline, month 6, month 12
  Intermetatarsal angle will be measured from the x-ray film taken in standing position with full weight bearing

SECONDARY OUTCOMES:
Change from baseline in pain score on 11-point Visual Analog Scale at month 3, month 6, month 9 and month 12 | Baseline, month 3, month 6, month 9 and month 12
  To measure the pain score of the hallux by using the numeric rating scale in the 3rd, 6th, 9th and 12th month

OTHER OUTCOMES:
Compliance of using Mold Making Silicone Toe Separator | Baseline, month 3, month 6, month 9 and month 12
  To identify the compliance by questionnaire in the 6th and 12th month, and self report (diary)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkok Noi, Bangkok, Thailand